CLINICAL TRIAL: NCT01144832
Title: IBS Treatment With H1-receptor Antagonists
Brief Title: Irritable Bowel Syndrome (IBS) Treatment With H1-receptor Antagonists
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S51638
Record Dates: First submitted 2010-05-28; First posted 2010-06-16 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: visceral hypersensitivity; mast cells
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ebastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo capsule (Placebo Comparator)
  Interventions: Drug: placebo capsule
- ebastine (Active Comparator)
  Interventions: Drug: ebastine

INTERVENTIONS:
Drug: ebastine — 20 milligram capsule once daily
  Arms: ebastine
Drug: placebo capsule — one capsule once daily
  Arms: placebo capsule

SUMMARY:
Purpose:

To evaluate the efficiency of Irritable Bowel Syndrome (IBS) patients treatment with the H1-receptor antagonist ebastine.

Design:

Double blind randomized placebo controlled trial. IBS patients receive a 12-weeks treatment with ebastine 20mg once daily or placebo (1:1 randomization).

End points:

End point is the effect of treatment on clinical symptoms and visceral hypersensitivity which will be evaluated with a barostat test.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome (ROME III criteria)
* age 18-65 years

Exclusion Criteria:

* medication: antidepressants or H1-receptor antagonists
* pregnancy, breast feeding
* co-morbidity: severe kidney- and/or liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on visceral sensitivity measured with rectal barostat. | after 12 weeks treatment

SECONDARY OUTCOMES:
Effect of treatment on IBS symptoms. | after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven
Locations (1):
- University hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Wouters MM, Balemans D, Van Wanrooy S, Dooley J, Cibert-Goton V, Alpizar YA, Valdez-Morales EE, Nasser Y, Van Veldhoven PP, Vanbrabant W, Van der Merwe S, Mols R, Ghesquiere B, Cirillo C, Kortekaas I, Carmeliet P, Peetermans WE, Vermeire S, Rutgeerts P, Augustijns P, Hellings PW, Belmans A, Vanner S, Bulmer DC, Talavera K, Vanden Berghe P, Liston A, Boeckxstaens GE. Histamine Receptor H1-Mediated Sensitization of TRPV1 Mediates Visceral Hypersensitivity and Symptoms in Patients With Irritable Bowel Syndrome. Gastroenterology. 2016 Apr;150(4):875-87.e9. doi: 10.1053/j.gastro.2015.12.034. Epub 2016 Jan 2. PMID 26752109